CLINICAL TRIAL: NCT00698165
Title: Observational Study on Costs and Caregiver Burden in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: i3 Innovus (Industry)
Responsible Party: Hans-Göran Hårdemark, Medical Science Director, AstraZeneca R&D
Other Study IDs: EHE 1100
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: 1200 adults with mild to severe Alzheimer's disease
- Caregivers: 1200 informal caregivers

SUMMARY:
Objective of study is to assess the costs of care, objective and subjective caregiver burden and quality of life in relation to disease severity measured by cognitive function, ADL capabilities and presence of behavioral disturbances in Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of possible or probable Alzheimer's disease, with or without vascular elements
* The primary caregiver can be identified
* The patient and his/her primary caregiver are both willing and able to participate in the study

Exclusion Criteria:

* Patient or caregiver affected by alcohol or narcotics to the extent that it interferes with the completion of the study
* Patient or caregiver does not understand English
* Patient and/ or caregiver is the physician or physician's staff
* Patient and/ or caregiver is a family member of the physician or physician's staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with Alzheimer's Disease and their informal caregivers are recruited from both outpatient settings and long-term residential care settings
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2007-06; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE), Disability Assessment for Dementia Scale (DAD), Neuropsychiatric Inventory Questionnaire (NPI-Q) | Collected one time only

SECONDARY OUTCOMES:
Resource Utilization in Dementia (RUD) | collected one time only
Short Form - 12 domains instrument (SF-12) | collected one time only
World Health Organization Quality of Life instrument (WHO-QoL) | collected one time only
Zarit Caregiver Burden Interview (ZBI) | collected one time only
15 domains Quality of Life Index instrument (15D) | collected one time only

CONTACTS AND LOCATIONS:
Overall Officials: Linus Jönsson, Study Director — i3 Innovus
Locations (82):
- United States (48):
  - Research Site, Northport, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Brentwood, California
  - Research Site, Fresno, California
  - Research Site, La Habra, California
  - Research Site, Long Beach, California
  - Research Site, Denver, Colorado
  - Research Site, Wetherfield, Connecticut
  - Research Site, Atlantis, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Tampa, Florida
  - Research Site, Titusville, Florida
  - Research Site, Venice, Florida
  - Research Site, Canton, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Belleville, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Prince Frederick, Maryland
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Eaton Rapids, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Eatontown, New Jersey
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Syracuse, New York
  - Research Site, Asheboro, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, East Providence, Rhode Island
  - Research Site, Beaufort, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Port Arthur, Texas
  - Research Site, Tyler, Texas
  - Research Site, Witchita Falls, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Gig Harbor, Washington
  - Research Site, Richland, Washington
- Spain (6):
  - Research Site, Cruces, Barakaldo
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Madrid
  - Research Site, Seville
- Sweden (13):
  - Research Site, Bergsjö
  - Research Site, Bromma
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Kristianstad
  - Research Site, Lomma
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Örnsköldsvik
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Varberg
- United Kingdom (15):
  - Research Site, Overton, Basingstoke
  - Research Site, Eastbourne, East Sussex
  - Research Site, Coney Hill, Gloucester
  - Research Site, Barnet, Hertfordshire
  - Research Site, Wood Green, London
  - Research Site, Brighton
  - Research Site, Chester
  - Research Site, Hove
  - Research Site, Ipswich
  - Research Site, Norwich
  - Research Site, Oxford
  - Research Site, Romsey
  - Research Site, Salisbury
  - Research Site, Stanmore
  - Research Site, Uckfield